CLINICAL TRIAL: NCT04028284
Title: Using Augmented Reality to 3D Map Needle Pathways in Real Time to Enhance Neuraxial Anesthesia
Brief Title: HoloLens: an Objective Alternative to the Operator's Memory
Acronym: Hololens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Fahad Alam, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Hololens
Record Dates: First submitted 2018-09-06; First posted 2019-07-22 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Virtual Reality; Anesthesia; Epidural
Keywords: epidural; analgesia; Virtual reality
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): In Group 1 (control), the staff anesthesiologist will follow the traditional technique for US-guided thoracic epidural insertion. Briefly, the anesthesiologist will use the US to identify and mark the appropriate spot for placement of the thoracic epidural catheter. The US probe is then placed at rest and the anesthesiologist will proceed with thoracic epidural needle insertion following standard techniques.
  Interventions: Other: US-guided epidural
- Group 2 (Active Comparator): In Group 2 (intervention), the staff anesthesiologist will use the HoloLens tool to assist with the traditional technique as described above for Group 1. In combination with the US, a hologram image of the trajectory towards the epidural space will be generated, thereby mitigating the need to walk off the lamina. The holographic system will mark the appropriate spot for placement of the thoracic epidural catheter. Then, the needle will be inserted following the holographic trajectory overlaid on the patient's back.
  Interventions: Device: HoloLens-guided epidural

INTERVENTIONS:
Device: HoloLens-guided epidural — To determine whether using the HoloLens tool increases the success of epidural insertion.
  Arms: Group 2
Other: US-guided epidural — traditional thoracic epidural procedure
  Arms: Group 1

SUMMARY:
Neuraxial anesthesia has traditionally been a 'blind' technique relying on users' feel and skill, both are subjective, lack complete accuracy and influenced by patient's physique variations that are quite challenging, and lead to patient morbidity, infection, and nerve injury. The ultrasound(US) use allows real-time views of needle position thereby achieving higher success rates, fewer complications, and reduced patient discomfort. While US guidance for neuraxial procedures is popular, it is still relatively uncommon due to technical and anatomical challenges. The study investigators have created an innovative methodology to use with HoloLens, an augmented reality tool, to provide an accurate live road map for the needle path hidden under the patient's skin. This see-through model is an objective alternative to the user's memory for direct visualization of the needle virtual trajectory as it passed through the tissue and towards the 3D printed bone. Also, this model may have a variety uses in anesthesia.

DETAILED DESCRIPTION:
US guidance for epidural anesthesia is yet challenging due to anatomical and technical restrictions which are rely on the operator's memory to imitate accurate needle trajectory. To address the problem, the study investigators designed and developed the first model of a live anatomical holographic marking system using Microsoft HoloLens, an augmented reality technology tool, to provide a superimposed US image as an objective alternative to the operator's memory. In this study, the proposed methodology will be used to accurate and ease directing the needle insertion thereby leading to the success of the epidural placement and decrease in procedure time. Based on previously published and data from the SHSC institution, mean thoracic epidural analgesia placement required 10 minutes with a standard deviation of 3 minutes. A reduction in procedure time will reduce patient discomfort, increase block and operating rooms efficiency thereby reducing hospital costs as well as used for anatomically challenging patients.

The investigators hypothesize that using augmented reality through HoloLens will lead to implementation of a newly developed virtual holographic 'see-through' tool for neuraxial anesthetic techniques that will increase needle accuracy and decrease procedure time.

The main question of the study is to assess the accuracy of the developed application. In particular, the study will determine if a holographic marking of the site of needle insertion and optimal angulation will increase needle accuracy and reduce procedure time by increasing first past success when compared to traditional ultrasound land-mark based techniques.

The methodology proposed in this study is truly innovative in medical content, involves a partnership with software and engineering experts. The study will lead to implementation of a new objective tool, validation of which will create an accessible, cost-effective piece of technology that will reduce patient morbidity and increase procedure success rate. This 'state-of-the-art' technology can be used for alternate procedures such as peripheral nerve block in patients that cannot be easily positioned for live US techniques. Also, this study will generate a knowledge-based approach that can be used as a teaching and clinical tool locally at institutions presented with anatomically difficult population (e.g. trauma, obstetric patients) at Sunnybrook Health Sciences Centre and around the world, where resources are at a minimum.

This is a prospective cohort randomized trial. With institutional ethical approval and having obtained both, written informed consent and verbal assent from participants, 84 thoracic epidural events will be assessed. A thoracic spine US 3D Phantom model utilizing open source BodyParts3D library anatomy files constructed by group of software and engineering experts, and accessible for practice to anesthetists. Our 3D Phantom model has similar palpation characteristics to a patient mimicking a standard loss of resistance to saline that occurs on entrance of a needle to the spinal canal cavity. The holographic mapping methodology will be practiced by anesthetists on the Phantom model until they feel comfortable with the system prior the study start. Participants will be recruited from the pre-anesthesia clinic. Only participants who meet inclusion criteria will be approached for participation in this study (Table 1,inclusion/exclusion criteria, study protocol). The anesthetists will be randomized to: Group1, landmark based thoracic epidural technique(control) or, Group 2, HoloLens-assisted thoracic epidural technique(intervention), where the needle will be inserted using instantly created holographic trajectory. SHS centre has a dedicated regional block room and four regional expert anesthetists in the US-guided thoracic epidural technique and are comfortable with the HoloLens. Prior to the study start, anesthetists will practice needle insertion on the phantom model by attempting needle insertion 20Xeach, or until they felt comfortable with the tool, while wearing HoloLens. Other aspects of patient care will follow the standard of care at the centre. Data will be collected by anesthetists and include patients surgical/abdominal pain assessment during epidural procedure and post-operatively, and questionnaire about their experience using the HoloLens.

Data will be validated to enable optimization and further implementation of novel technology.

1. Inclusion Criteria/Anesthetists:

   * Trained in US-guided epidural technique with fellowship
   * Performed >100 thoracic US-guided epidural procedures
2. Exclusion Criteria/Patients:

   * age >18
   * Lack of verbal patient assent after study introduction

The control group will be required to determine if hologram mapping and methodology indeed provide an accuracy of the holographic trajectory and create a live road map for the needle path hidden under the patient's skin. Study participants will be withdrawn from the study at their request at any time.

To address this study specific objectives of whether the HoloLens application, that is designed to allow a holographic marking of the needle insertion site and optimal angulation would 1) decrease procedure time by increasing first past success when used as a guide to the thoracic epidural space; and 2) increase needle accuracy when compared to traditional ultrasound landmark based techniques, an observer (i.e. anesthesiologist) will document following:

1. the time to procedure completion starting from skin puncture to time at which the Tuohy needle is withdrawn;
2. the number of a needle movements (in any direction/re-direction)
3. number of skin punctures made;
4. patients' pain score during the procedure and post-operatively using the numeric rating scale (NRS);
5. any complications during the procedure such as paresthesias, dural punctures;
6. the need for patient controlled analgesia (PCA) in PACU (constituting failure of epidural).

ELIGIBILITY:
Inclusion Criteria:

* Trained in US-guided epidural technique with fellowship
* Performed >100 thoracic US-guided epidural procedures

Exclusion Criteria:

* Age <18
* Lack of verbal patient assent after study introduction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wiegelmann J, Choi S, McHardy PG, Matava C, Singer O, Kaustov L, Alam F. Randomized control trial of a holographic needle guidance technique for thoracic epidural placement. Reg Anesth Pain Med. 2024 Dec 2;49(12):861-866. doi: 10.1136/rapm-2023-104703. PMID 38212048
- [Derived] Tanwani J, Alam F, Matava C, Choi S, McHardy P, Singer O, Cheong G, Wiegelmann J. Development of a Head-Mounted Holographic Needle Guidance System for Enhanced Ultrasound-Guided Neuraxial Anesthesia: System Development and Observational Evaluation. JMIR Form Res. 2022 Jun 23;6(6):e36931. doi: 10.2196/36931. PMID 35737430

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant was not randomized due to their surgery being cancelled.
Groups:
- Group C: In Group C (control), the staff anesthesiologist will follow the traditional technique for US-guided thoracic epidural insertion. Briefly, the anesthesiologist will use the US to identify and mark the appropriate spot for placement of the thoracic epidural catheter. The US probe is then placed at rest and the anesthesiologist will proceed with thoracic epidural needle insertion following standard techniques.
  US-guided epidural: traditional thoracic epidural procedure
- Group H: In Group H (intervention), the staff anesthesiologist will use the HoloLens tool to assist with the traditional technique as described for Group C. In combination with the US, a hologram image of the trajectory towards the epidural space will be generated, thereby mitigating the need to walk off the lamina. The holographic system will mark the appropriate spot for placement of the thoracic epidural catheter. Then, the needle will be inserted following the holographic trajectory overlaid on the patient's back.
  HoloLens-guided epidural: To determine whether using the HoloLens tool increases the success of epidural insertion.
Period: Overall Study
Arm/Group | Group C | Group H
Started | 42 | 41
Completed | 42 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group C | Group H | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (14.2) | 62.9 (13.3) | 64.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 22 | 22 | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Surgical Type [Count of Participants; unit: Participants]
  General | 3 | 3 | 6
  Gynecologic | 10 | 13 | 23
  Oncology | 25 | 24 | 49
  Urologic | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Procedure Time
Description: The time starting from skin puncture until withdrawal of the Tuohy needle after successful catheter placement.
Time Frame: During procedure
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group C | Group H
Number analyzed (Participants) | 42 | 41
Minutes | 7.3 (6.0) | 4.5 (4.6)
Statistical Analysis 1: Comparison: Group C vs Group H; Test type: Other — Two-sided inferential test; p = 0.02, t-test, 2 sided — Adjusted for multiple comparisons using the Holm-Bonferroni correction. The a priori threshold for statistical significance was P < 0.05 for the primary outcome

2. Secondary Outcome: Number of Needle Insertions
Description: The number of times the needle was completely withdrawn from the skin and reinserted at a new location.
Time Frame: During procedure
Measure: Mean (Standard Deviation); unit: Insertions
Arm/Group | Group C | Group H
Number analyzed (Participants) | 42 | 41
Insertions | 1.5 (1.0) | 1.3 (0.5)
Statistical Analysis 1: Comparison: Group C vs Group H; Test type: Other — Inferential two-sided test; p = 0.31, t-test, 2 sided

3. Secondary Outcome: Number of Needle Passes
Description: Any advancement of of the needle along an unchanged trajectory.
Time Frame: During procedure
Measure: Mean (Standard Deviation); unit: Number of passes
Arm/Group | Group C | Group H
Number analyzed (Participants) | 42 | 41
Number of passes | 14.4 (16.3) | 7.2 (7.9)
Statistical Analysis 1: Comparison: Group C vs Group H; Test type: Other — Inferential two-sided test; p = 0.01, t-test, 2 sided — Adjusted for multiple comparisons using the Holm-Bonferroni correction

4. Secondary Outcome: Number of Bone Contacts
Description: The number of times the needle contacted a bone, as reported by the anesthesiologist performing the procedure.
Time Frame: During procedure
Measure: Mean (Standard Deviation); unit: Number of contacts
Arm/Group | Group C | Group H
Number analyzed (Participants) | 42 | 41
Number of contacts | 12.2 (16) | 6 (8.0)
Statistical Analysis 1: Comparison: Group C vs Group H; Test type: Other — Inferential two-sided test; p = 0.03, t-test, 2 sided — Adjusted for multiple comparisons using the Holm-Bonferroni correction

5. Secondary Outcome: Procedural Pain
Description: Procedural pain assessed using the numerical rating scale (0-10, with 0 indicating no pain and 10 the worst possible pain) after the completion of the epidural procedure.
Time Frame: During procedure
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group C | Group H
Number analyzed (Participants) | 42 | 41
Units on a scale | 2.6 (1.6) | 2.8 (2.3)
Statistical Analysis 1: Comparison: Group C vs Group H; Test type: Other — Inferential two-sided test; p = 0.56, t-test, 2 sided

6. Secondary Outcome: Pain in PACU
Description: Pain assessed using the numerical rating scale (0-10, with 0 indicating no pain and 10 the worst possible pain) in the post-anesthesia care unit.
Time Frame: In the PACU
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group C | Group H
Number analyzed (Participants) | 42 | 41
Units on a scale | 2.6 (3.0) | 2.4 (2.8)
Statistical Analysis 1: Comparison: Group C vs Group H; Test type: Other — Inferential two-sided test; p = 0.78, t-test, 2 sided

7. Secondary Outcome: Number of Participants With Epidural Failure
Description: Defined as unexpected addition of intravenous patient controlled analgesia to the patient's pain control regimen prior to discharge from the recovery room.
Time Frame: In the PACU
Measure: Count of Participants; unit: Participants
Arm/Group | Group C | Group H
Number analyzed (Participants) | 42 | 41
Participants | 3 | 0
Statistical Analysis 1: Comparison: Group C vs Group H; Test type: Other — Inferential two-sided test; p = 0.24, Fisher Exact

8. Secondary Outcome: Complications
Description: Complications such as paresthesia and dural puncture as noted by the observer.
Time Frame: During procedure
Measure: Number; unit: Number of complications
Arm/Group | Group C | Group H
Number analyzed (Participants) | 42 | 41
Number of complications | 0 | 0

ADVERSE EVENTS:
Time Frame: During the procedure.
Arm/Group | Group C | Group H
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41
Other Adverse Events (participants affected / at risk) | 0/42 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT04028284/Prot_SAP_000.pdf